CLINICAL TRIAL: NCT02381600
Title: An Evaluation of the Effects of Vitamin D Supplementation on Specific Cognitive Functions and Depressive Symptoms of Older Subjects With Low Levels of This Vitamin
Brief Title: An Evaluation of the Effect of Vitamin D Supplementation on the Cognitive Function of Older Subjects With Low Levels of This Vitamin
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulties recruiting participant
Sponsor: Meir Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ק096/2014
Record Dates: First submitted 2015-02-08; First posted 2015-03-06 (Estimated); Last update posted 2021-02-25 (Actual); Status verified 2016-10

CONDITIONS: VITAMIN D DEFICIENCY
Keywords: vitamin D; aging; cognitive function; depression; executive function
MeSH Terms: conditions — Vitamin D Deficiency; Depression | interventions — Vitamin D

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Intervention group- vitamin D (Experimental): Include patients aged 65 years and older that are found to have below-normal serum levels of vitamin D on routine laboratory testing. After providing informed consent (the study was submitted for approval by the Ethics Committee of the Clalit Health Services) eligible subjects will undergo cognitive and affective assessment
  Interventions: Drug: Vitamin D

INTERVENTIONS:
Drug: Vitamin D — Experimental :
  1. Patients will undergo clinical and functional assessment as well as evaluation using the Montreal Cognitive Assessment (MoCA) screening test, the modified 15-item Geriatric Depression Scale, and the Neurotrax (®Mindstreams) computerised cognitive assessment battery.
  2. Patients will receive a supplemental monthly oral dose of 60000 units Vitamin D administered by a nurse for a period of 3 months Patients will undergo a repeat blood test to examine the level of vitamin D at the end of 3 months of follow-up.
  3. At 3-month follow-up atients will be asked to complete the 15-item GDS and the Neurotrax (®Mindstreams) computerised cognitive assessment battery.

SUMMARY:
Background: Ageing is associated with an increased risk of cognitive decline and depression. Vitamin D plays an important role in many of the symptoms and conditions related to advanced age, including impaired balance, falls and osteoporosis. Vitamin D also has a physiological effect on the function of the central nervous system, and studies have suggested a relationship between this vitamin and changes in affect and cognitive function in the elderly. The investigators propose a pilot study to examine the relationship between below-normal levels of Vitamin D to affective symptoms and specific cognitive functions in the elderly.

Methods: A total of 30 subjects of both genders older than 65 years with levels of 25-OH Vitamin D lower than 30 ng/ml on routine laboratory screening will be referred by the treating family physicianfor screening. Subjects will be required to provide written informed consent for inclusion in the study. Exclusion criteria will include any active or unstable medical condition as determined by the treating physician, known neurocognitive disorder, known affective disorder, the use of any class of antidepressant drugs, the use of supplements containing vitamin D in any dose, significant visual or hearing impairment not corrected by spectacles or hearing aids, and a level of literacy that limits cognitive ability. All subjects will undergo cognitive screening by use of the MoCA test, computerized cognitive assessment using the the Neurotrax (®Mindstreams) computerised cognitive assessment battery, and the 15-item Geriatric Depression Scale. All subjects will undergo repeat testing for level of 25-OH Vitamin D, and where below-normal levels are confirmed patients will receive a supplemental monthly oral dose of 60000 units Vitamin D administered by a nurse for a period of 3 months. At 3 months subjects will undergo repeat testing for level of 25-OH Vitamin D, and repeat computerized cognitive assessment using the Neurotrax Mindstreams battery and the 15-item Geriatric Depression Scale (GDS).

DETAILED DESCRIPTION:
Background: Ageing is associated with an increased risk of cognitive decline and depression. Vitamin D plays an important role in many of the symptoms and conditions related to advanced age, including impaired balance, falls and osteoporosis. Vitamin D also has a physiological effect on the function of the central nervous system, and studies have suggested a relationship between this vitamin and changes in affect and cognitive function in the elderly. The investigators propose a pilot study to examine the relationship between below-normal levels of Vitamin D to affective symptoms and specific cognitive functions in the elderly.

Methods: A total of 30 subjects of both genders older than 65 years with levels of 25-OH Vitamin D lower than 30 ng/ml on routine laboratory screening will be referred by the treating family physicianfor screening. Subjects will be required to provide written informed consent for inclusion in the study. Exclusion criteria will include any active or unstable medical condition as determined by the treating physician, known neurocognitive disorder, known affective disorder, the use of any class of antidepressant drugs, the use of supplements containing vitamin D in any dose, significant visual or hearing impairment not corrected by spectacles or hearing aids, and a level of literacy that limits cognitive ability. All subjects will undergo cognitive screening by use of the MoCA test, computerized cognitive assessment using the the Neurotrax (®Mindstreams) computerised cognitive assessment battery, and the 15-item Geriatric Depression Scale. All subjects will undergo repeat testing for level of 25-OH Vitamin D, and where below-normal levels are confirmed patients will receive a supplemental monthly oral dose of 60000 units Vitamin D administered by a nurse for a period of 3 months. At 3 months subjects will undergo repeat testing for level of 25-OH Vitamin D, and repeat computerized cognitive assessment using the Neurotrax Mindstreams battery and the 15-item Geriatric Depression Scale (GDS).

Study Type: An open-label prospective pilot interventional study

Study Design: the one group pretest-posttest design.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 65 years and older.
* Level of vitamin D (25-OH vitamin D) is less than 30 ng / ml.
* Stable health status as assessed by the treating primary care physician.
* Do not take antidepressant medications.
* Do not take supplements containing vitamin D.
* Normal cognitive function as determined by MoCA Test screening and clinical assessment
* Adequate literacy to enable the performance of assessment instruments
* Provide informed consent as required by the Ethics Committee.

Exclusion Criteria:

* Age younger than 65 years
* Health status not stable as determined by the treating primary care physician
* Cognitive impairment or dementia
* Illiteracy
* Taking supplements containing Vitamin D
* Taking antidepressant medications
* Significant visual or hearing impairment not corrected by spectacles or hearing aids
* Impaired competency limiting the subject's ability to provide informed consent

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 1 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Cognitive function as assessed by the Neurotrax (®Mindstreams) computerised cognitive assessment battery | Baseline and 3-month follow-up
  Change in cognitive function at 3 months compared to baseline according to cognitive indices on a computerized assessment battery

CONTACTS AND LOCATIONS:
Locations (1):
- Yan Press, Beersheba, Israel